CLINICAL TRIAL: NCT03124641
Title: Hypothermic Oxygenated Machine Perfusion (HOPE) for Liver Transplantation of Human Liver Allografts From Extended Criteria Donors (ECD) in Donation After Brain Death (DBD); a Multicenter Randomized Controlled Trial (HOPE ECD-DBD)
Brief Title: HOPE for Human Extended Criteria and Donation After Brain Death Donor (ECD-DBD) Liver Allografts
Acronym: HOPE-ECD-DBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Aachen (Other)
Responsible Party: Principal Investigator, Georg Lurje, M.D., Attending Transplant Surgeon, University Hospital, Aachen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 049/17
Record Dates: First submitted 2017-03-20; First posted 2017-04-24 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Injury; Liver Transplant
Keywords: Hypothermic oxygenated machine perfusion; Orthotopic liver transplantation; Extended criteria donation; Donation after brain death; HOPE

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic oxygenated perfusion (HOPE) (Experimental): Application of Hypothermic machine perfusion (HOPE) for 1-2 hours
  Interventions: Device: Hypothermic oxygenated perfusion (HOPE)
- Conventional cold storage (CCS) (Active Comparator): Conventional cold storage
  Interventions: Procedure: Conventional cold storage (CCS)

INTERVENTIONS:
Device: Hypothermic oxygenated perfusion (HOPE) — HOPE for 1 hour via the portal vein in a recirculating and pressure controlled system (2-3 mm Hg), 0.1 ml/g liver/min, perfusion volume 3-4 L, Belzer (UW) machine perfusion solution, perfusate temperature 10 °C, perfusate oxygenation pO2 of 60-80 kPa
  Other Names: Hypothermic machine perfusion (HMP)
  Arms: Hypothermic oxygenated perfusion (HOPE)
Procedure: Conventional cold storage (CCS) — Conventional static cold storage (CCS) on temperature 4-6 °C from organ procurement
  Other Names: CCS
  Arms: Conventional cold storage (CCS)

SUMMARY:
The purpose of this study is to test the effects of hypothermic oxygenated machine perfusion (HOPE) in a phase-II prospective multicenter randomized clinical trial (RCT) on extended criteria donor allografts (ECD) in donation after brain death (DBD) orthotropic liver-transplantation (OLT) (HOPE-ECD-DBD). Human whole organ liver grafts will be submitted to 1-2 hours of HOPE via the portal vein directly before implantation and going to be compared to a control-group of patients transplanted after conventional cold storage (CCS). Primary (early graft injury) and secondary (e.g. postoperative complications, hospital stay, survival) objectives are going to be analysed in a 12 month follow up. Ischemia-reperfusion (I/R) injury and inflammation will be assessed using liver tissue, serum and bile samples as well as machine perfusion perfusate.

To improve the availability of donor allografts and reduce waiting list mortality, graft acceptance criteria were extended increasingly over the decades. The use of extended criteria donor (ECD) allografts is associated with higher incidences of primary graft non-function (PNF) and/or delayed graft function (DGF). As such, several strategies have been developed aiming at "reconditioning" poor quality ECD grafts. HOPE has been tested intensively in pre-clinical animal experiments. Although, its known that HOPE can exert its reconditioning effect via cellular and mitochondrial pathways in the endothelial and parenchymal cells, there is still scarce evidence available on the exact subcellular mechanism of HOPE induced organ protection in the clinical scenario of liver transplantation. In donation after cardiac death (DCD) OLT, the positive effects of HOPE have been shown to reduce the incidence of biliary complications, mitochondrial damage and improve the overall cellular energy-status.

In the HOPE setting, organ perfusion is performed in the transplant center shortly before the actual implantation with oxygenated perfusate using an extra corporal organ perfusion system. The first clinical study with this promising technique was recently reported in a Swiss cohort of patients who received DCD allografts. In organ donation after brain death (DBD), the only legally accepted approach for organ donation in most countries, HOPE and its effect on early graft injury and postoperative complications remains to be elucidated.

DETAILED DESCRIPTION:
The present RCT comprises two groups, a perfusion (group 1; HOPE) and a control conventional cold storage (group 2; CCS) group. Patients with proven written informed consent on waiting list for orthotopic liver transplantation will be recruited. Randomization is performed with an online randomizing tool for clinical trials (www.randomizer.at) at the time of allograft arrival at the transplant center and acceptance of the organ for transplantation. Stratified randomization model will be used to ensure balance of prognostic variables between the treatment groups.

In case of randomisation to group 1, HOPE will be applied to the allograft in the operation room, directly after the back table preparation. The application of HOPE to the liver allograft will not delay the implantation due to the fact that it is performed parallel to the recipient hepatectomy.

Commercially available and machine-perfusion approved Belzer MPS® UW solution (Belzer Organ Preservation Solutions, Bridge for Life) will be used as perfusate for machine perfusion.

Patients will be followed for one year after OLT.

Interim analysis: After n=12 per randomized group is reached, data will be analyzed by an independent Data Monitoring Committee. The RCT will be stopped if one of the following criteria is reached:

Significantly higher serum ALT levels (p<0.001 using Student's t-test) in the HOPE group compared to the CCS group (Efficacy).

The proportion of Grade ≥ III complications is significantly higher (p<0.05, Fischer's exact test) in the HOPE group when compared to the CCS group (Safety).

ELIGIBILITY:
Inclusion Criteria:

-Patients with signed informed consent, suffering from end stage-liver disease and/or malignant liver tumors listed for liver transplantation and receiving ECD organs.

ECD Criteria are defined as:

* Donors 65 years of age and older
* Intensive therapy of the donor was required before donation for at least 7 days, --Obesity of the donor with a Body Mass Index > 30
* Fatty liver (with histology) > 40 %
* Serum-Sodium > 165 mmol/l
* Serum AST or ALT > 3 x normal, Serum-Bilirubin > 2 mg/dl)

Exclusion Criteria:

* Recipients of split of living donor liver transplants
* Previous liver transplantation
* Combined transplantations (liver-kidney, liver-lung, etc.)
* Participation in other liver related trials
* The subject received an investigational drug within 30 days prior to inclusion
* The subject is unwilling or unable to follow the procedures outlined in the protocol
* The subject is mentally or legally incapacitated
* Patient is not able to understand the procedures due to language barriers
* Family members of the investigators or employees of the participating department

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Early graft injury | During the first week postoperatively (absolute and relative delta)
  Peak serum alanine aminotransferase-ALT

SECONDARY OUTCOMES:
Postoperative complications | Subjects will be followed for one year postoperatively
  Clavien-Dindo complication score
Cumulative postoperative complications | Subjects will be followed for one year postoperatively
  Comprehensive complication index (CCI)
Early allograft dysfunction (EAD) | During the first week postoperatively
  Olthoff criteria (bilirubin 10mg/dL on day 7, international normalized ratio 1.6 on day 7, and alanine or aspartate aminotransferases >2000 IU/L)
Duration of intensive care stay | Subjects will be followed for one year postoperatively
  Duration of ICU stay
Duration of hospital stay | Subjects will be followed for one year postoperatively
  Duration of hospitalisation
One-year recipient- and graft survival | Subjects will be followed for one year postoperatively
  One year patient and graft survival
Ischemia-reperfusion injury and inflammatory responses | Before preservation (HOPE or CCS), after liver implantation (0-3 hrs)
  Liver samples taken upon arrival of the organ (before HOPE or corresponding cold-storage), and at the end of the implantation procedure before closure of the abdomen
(in selected centers) Biliary epithelial cell injury | Postoperative days 1, 2, and 3
  Bile samples collected from T-Drain

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lurje, M.D., Principal Investigator — RWTH Aachen University I Charité-Universitätsmedizin Berlin
Locations (4):
- Department of Transplantation Surgery, Institute for Clinical and Experimental Medicine, Prague, Czechia
- Germany (3):
  - Department of Surgery and Transplantation, University Hospital RWTH Aachen, Aachen
  - Department of Surgery, Campus Charité Mitte | Campus Virchow-Klinikum, Charité-Universitätsmedizin Berlin, Germany, Berlin
  - Department of General, Visceral, and Transplant Surgery, Ludwig-Maximilians-University Munich, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czigany Z, Schoning W, Ulmer TF, Bednarsch J, Amygdalos I, Cramer T, Rogiers X, Popescu I, Botea F, Fronek J, Kroy D, Koch A, Tacke F, Trautwein C, Tolba RH, Hein M, Koek GH, Dejong CHC, Neumann UP, Lurje G. Hypothermic oxygenated machine perfusion (HOPE) for orthotopic liver transplantation of human liver allografts from extended criteria donors (ECD) in donation after brain death (DBD): a prospective multicentre randomised controlled trial (HOPE ECD-DBD). BMJ Open. 2017 Oct 10;7(10):e017558. doi: 10.1136/bmjopen-2017-017558. PMID 29018070
- [Derived] Schliephake F, Lurje I, Uluk D, Eden J, Czigany Z, Pein J, Husen P, Engelmann C, Michalski C, Kohlhepp M, Strnad P, Dutkowski P, Tacke F, Neumann UP, Meierhofer D, Lurje G. Effects of hypothermic oxygenated machine perfusion on bile composition after liver transplantation - Findings from a randomized controlled trial. JHEP Rep. 2025 Oct 17;8(2):101647. doi: 10.1016/j.jhepr.2025.101647. eCollection 2026 Feb. PMID 41551407
- [Derived] Czigany Z, Pratschke J, Fronek J, Guba M, Schoning W, Raptis DA, Andrassy J, Kramer M, Strnad P, Tolba RH, Liu W, Keller T, Miller H, Pavicevic S, Uluk D, Kocik M, Lurje I, Trautwein C, Mehrabi A, Popescu I, Vondran FWR, Ju C, Tacke F, Neumann UP, Lurje G. Hypothermic Oxygenated Machine Perfusion Reduces Early Allograft Injury and Improves Post-transplant Outcomes in Extended Criteria Donation Liver Transplantation From Donation After Brain Death: Results From a Multicenter Randomized Controlled Trial (HOPE ECD-DBD). Ann Surg. 2021 Nov 1;274(5):705-712. doi: 10.1097/SLA.0000000000005110. PMID 34334635
- See also: HOPE ECD-DBD webpage — http://www.hopeliver.com